CLINICAL TRIAL: NCT01503294
Title: Comparison of Temporal to Pulmonary Artery Temperature Measurement in Patients With Fever
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Diane L. Carroll, Principal Investigator, Massachusetts General Hospital
Other Study IDs: TAT-1
Record Dates: First submitted 2011-12-30; First posted 2012-01-04 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Fever
Keywords: Temporal artery thermometer; Pulmonary artery thermistor
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Assessment and evaluation of body temperature is an important sign of health and disease. Inferior thermometry increases the risk of morbidity and mortality, and increases health care cost by delaying the diagnosis and treatment of fever-related disease. The gold standard for measuring core body temperature is the pulmonary artery thermistor (PAT). The measurement of the PAT requires the insertion of the invasive pulmonary artery catheter, a high risk procedure.

An innovative thermometry technology, the temporal artery thermometer (TAT), has been introduced into the clinical arena as a potential non-invasive proxy for the PAT. The TAT reduces the risk and cost of pulmonary artery catheter insertion by non-invasively measuring core blood temperature by measuring temperature over the skin of the temporal artery.

Research to demonstrate the precision and accuracy of the TAT in normothermic patients has been published, but little to no data is available in those with temperatures greater than 100.4oF. The purpose of this study is to measure the precision and accuracy of 2standard of care temperature methods: the thermistor from the PAT, considered the gold standard, and the TAT as measured in those patients with a PAT temperature greater than 100.4oF.

DETAILED DESCRIPTION:
The results from previous studies agree that direct comparisons of the PAT and TAT are clinically comparable in the normal temperature range in adults. This was defined as a clinical significance difference of less than ±.5ºC (.9ºF. In the one study that assessed subjects with fevers (temperatures greater than 37.8oC (100.0oF) with some methodological criticism, compared the TAT to PAT in adults (n=15). There were poor correlations (r=0.3) among the adult measurements with a difference of 1.3+0.6o C. Eighty-nine percent of the TAT measurements were different than the PAT by more that ±.5ºC.

With only one study that focused in those who had a PAT outside the normal temperature range to evaluate accuracy and precision, there is a need for further research to assess the accuracy and precision of the TAT for detection of hyperthermia. A new onset of temperature equal to or above 100.4oF is defined as a fever and a temperature of 100.9oF is considered a reasonable trigger for a clinical assessment according to the Society of Critical Care Medicine in their fever guidelines for adults. Researchers synthesizing the literature on the TAT and other noninvasive temperature measurements, indicate that noninvasive temperature measurements are accurate for normal temperatures but may fail to detect hyperthermia and hypothermia, depending on the thermometer used. The authors concluded that the TAT is clinically comparable to the PAT in only the normal temperature range.

A repeated measures design will be used to describe the accuracy and precision of 2 temperature measurements, the PAT and the TAT. Study subjects will act as their own control in order to investigate the difference in PAT readings and the TAT readings in both the core and oral mode. The PAT will also be compared to the TAT reading taken by the clinical staff.

ELIGIBILITY:
Inclusion Criteria:

1. Pulmonary artery catheter in place for a clinical indication,
2. fever > 100.4oF

Exclusion Criteria:

1. significant carotid or cerebrovascular disease,
2. PA catheter is not in proper position as confirmed by chest x-ray

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
accuracy and precision of the TAT as compared to the PAT | 1 minute
  Recorded temperature from the PAT and then collected TAT temperature.

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Carroll, PhD, RN, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States